CLINICAL TRIAL: NCT03560739
Title: A 12 Week Randomized Open Label Parallel Group Multicenter Study to Evaluate Bioequivalence of 20 mg Subcutaneous Ofatumumab Injected by Pre-filled Syringe or Autoinjector in Adult RMS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157G2102
Record Dates: First submitted 2018-05-15; First posted 2018-06-18 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; Relapsing-remitting Multiple Sclerosis; Secondary progressive Multiple Sclerosis; Bioequivalence; Pharmacokinetics; Neurofilament light chain; Pre-filled Syringe; Auto-injector; adult; AI; PFS; OMB157
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Charcot-Marie-Tooth disease, Type 1F | interventions — ofatumumab; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: To address the primary objective of testing bioequivalence at dosing interval after Week 8 between Pre-filled Syringe (PFS) and Auto-Injector (AI), the primary analysis involves the two groups (PFS (abdomen) and AI (abdomen)). Further the pharmacokinetcs of ofatumumab will be compared between using the thigh or abdomen for injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OMB 20mg PFS abdomen (Other): ofatumumab 20 mg subcutaneous (sc.) injection with pre-filled syringes (PFS) administrated on abdomen
  Interventions: Combination Product: ofatumumab with PRF
- OMB 20mg AI abdomen (Other): ofatumumab 20 mg subcutaneous (sc.) injection with autoinjector (AI) administrated on abdomen
  Interventions: Combination Product: ofatumumab with AI
- OMB 20mg PFS thigh (Other): ofatumumab 20 mg subcutaneous (sc.) injection with pre-filled syringes (PFS) administrated on thigh
  Interventions: Combination Product: ofatumumab with PRF
- OMB 20mg AI thigh (Other): ofatumumab 20 mg subcutaneous (sc.) injection with autoinjector (AI) administrated on thigh
  Interventions: Combination Product: ofatumumab with AI

INTERVENTIONS:
Combination Product: ofatumumab with PRF — ofatumumab 20 mg subcutanious injection administered with pre-filled syringe (PRF)
  Arms: OMB 20mg PFS abdomen; OMB 20mg PFS thigh
Combination Product: ofatumumab with AI — ofatumumab 20 mg subcutaneous injection administered with autoinjector (AI)
  Arms: OMB 20mg AI abdomen; OMB 20mg AI thigh

SUMMARY:
The primary purpose of this study is to demonstrate pharmacokinetic bioequivalence of ofatumumab injected by Pre-filled Syringe (PFS) versus Auto-Injector (AI) devices and thereby establish a bridge between the ongoing Phase 3 program and the to-be-marketed drug-device combinations

DETAILED DESCRIPTION:
Characterization of the pharmacokinetics of ofatumumab administered via the PFS used inclinical trials and the to-be-marketed autoinjector at the clinical dose of 20 mg will be conducted after an initial depletion of CD20 positive B-cells. Comparing the ofatumumab pharmacokinetics between the two drug-device combinations only after the induction period is expected to reduce initial high variability due to target-mediated clearance. This ensures a more stable baseline for PK comparison in a parallel group study design and reflects the clinical situation where systemic concentrations are at steady-state. In order to justify the resulting longterm B-cell depletion, a PK comparability study between the PFS and the AI can only be conducted in MS patients rather than in healthy subjects to balance the risk/benefit and to obtain PK data from the relevant patient population. In order for patients to obtain a clinical benefit from participation in the study, continued treatment with ofatumumab will be offered to all eligible patients through enrollment into the open-label Phase 3 extension study (separate protocol, COMB157G2399).

A secondary objective of the study is to characterize the pharmacokinetics following subcutaneous administration of ofatumumab to either the abdominal region or the thigh which are two injections sites allowed in the Phase 3 study and planned for inclusion in the label. Another secondary objective is assessment of immunogenicity during the 12 weeks duration of the study addressing potential differences in ofatumumab anti-drug antibody formation between the PFS and AI devices as well as between abdomen and thigh injection sites.

This was a randomized, open-label, multi-center, parallel group 12-week study to evaluate the pharmacokinetic bioequivalence of ofatumumab injected by pre-filled syringe (PFS) or autoinjector (AI) devices. The study design included four parallel groups of relapsing multiple sclerosis (RMS) patients. Assessment of the primary and secondary endpoints was based on data collected through the dosing interval between Week 8 and Week 12 where approximate steady-state pharmacokinetics was anticipated.

All patients received open-label ofatumumab 20 mg sc every 4 weeks (after an initial loading regimen of three weekly 20 mg doses in the first 14 days) and were randomized (5:5:1:1) into 4 groups dependent on device and location of injection. Randomization was not blinded. Groups: 1: PFS, abdomen, 2: AI, abdomen 3: PFS, thigh 4: AI, thigh.

The study had 3 Parts. Part 1 was a 30 day screening period. Part 2 was a treatment period which had an induction period of 4 weeks, followed by 4 weeks to ensure steady state was reached and a 4 week pharmacokinetics phase for a total of 12 weeks.

Part 3 was a safety follow-up period for patients who completed the study but did not enter the extension study and patients who prematurely discontinued the study. This period was 9 months for patients who had repleted their B-cells (back to baseline value). For patients who had not repleted their B-cells, 3 month assessments were done until their B-cells were repleted or patients had initiated other disease modifying/immunosuppressive thereapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (MS)
* Relapsing MS: relapsing-remitting course (RRMS), or Secondary progressive (SPMS) course
* EDSS score of 0 to 5.5
* Documentation of at least: 1 relapse during the previous year OR 2 relapses during the previous 2 years prior to Screening OR a positive Gd-enhancing MRI scan during the year prior to randomization.
* Neurologically stable within 1 month prior to randomization

Exclusion Criteria:

* Patients with primary progressive MS or SPMS without disease activity
* Disease duration of more than 10 years in patients with EDSS score of 2 or less
* Patients with an active chronic disease of the immune system other than MS
* Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS or to test positive for HIV antibody at Screening
* Patients with neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML), or confirmed PML

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (12):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Basalt, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Ozark, Missouri
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, Sherman, Texas
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Sofia, Bulgaria
- Czechia (5):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Havířov, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Pardubice
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Castilleja de la Cuesta, Sevilla

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bar-Or A, Montalban X, Hu X, Kropshofer H, Kukkaro P, Coello N, Ludwig I, Willi R, Zalesak M, Ramanathan K, Kieseier BC, Haring DA, Bagger M, Fox E. Serum Neurofilament Light Trajectories and Their Relation to Subclinical Radiological Disease Activity in Relapsing Multiple Sclerosis Patients in the APLIOS Trial. Neurol Ther. 2023 Feb;12(1):303-317. doi: 10.1007/s40120-022-00427-8. Epub 2022 Dec 19. PMID 36534274
- [Derived] Jones B, Li B, Bagger M, Goodyear A, Ludwig I. Statistical methodology for highly variable compounds: A novel design approach for the ofatumumab Phase 2 bioequivalence study. Pharm Stat. 2022 Nov;21(6):1357-1365. doi: 10.1002/pst.2233. Epub 2022 May 23. PMID 35604539
- [Derived] Bar-Or A, Wiendl H, Montalban X, Alvarez E, Davydovskaya M, Delgado SR, Evdoshenko EP, Giedraitiene N, Gross-Paju K, Haldre S, Herrman CE, Izquierdo G, Karelis G, Leutmezer F, Mares M, Meca-Lallana JE, Mickeviciene D, Nicholas J, Robertson DS, Sazonov DV, Sharlin K, Sundaram B, Totolyan N, Vachova M, Valis M, Bagger M, Haring DA, Ludwig I, Willi R, Zalesak M, Su W, Merschhemke M, Fox EJ. Rapid and sustained B-cell depletion with subcutaneous ofatumumab in relapsing multiple sclerosis: APLIOS, a randomized phase-2 study. Mult Scler. 2022 May;28(6):910-924. doi: 10.1177/13524585211044479. Epub 2021 Oct 4. PMID 34605319
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=715

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 344 participants were screened
Groups:
- OMB 20mg AI Abdomen: Ofatumumab 20 mg subcutaneous (s.c.) injection with autoinjector (AI) administrated on abdomen
- OMB 20mg PFS Abdomen: Ofatumumab 20 mg subcutaneous (s.c.) injection with pre-filled syringes (PFS) administrated on abdomen
- OMB 20mg AI Thigh: Ofatumumab 20 mg subcutaneous (s.c.) injection with autoinjector (AI) administrated on thigh
- OMB 20mg PFS Thigh: Ofatumumab 20 mg subcutaneous (s.c.) injection with pre-filled syringes (PFS) administrated on thigh
Period: Overall Study
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh
Started | 128 | 130 | 13 | 13
Completed | 128 | 129 | 13 | 13
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh | Total
Number analyzed (Participants) | 128 | 130 | 13 | 13 | 284
Age, Customized [Number; unit: participants]
  18 to 30 years | 32 | 29 | 5 | 2 | 68
  31 to 40 years | 42 | 53 | 3 | 10 | 108
  41 to 55 years | 54 | 48 | 5 | 1 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 90 | 9 | 8 | 199
  Male | 36 | 40 | 4 | 5 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 4 | 0 | 0 | 6
  White | 125 | 125 | 13 | 12 | 275
  Mixed | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence of 20 mg Ofatumumab Injected by Pre-filled Syringe (PFS) vs Autoinjector (AI) to Abdomen as Measured by AUCtau
Description: Bioequivalence of AUCtau ) will be measured over the time period of Week 8 to Week 12 dosing interval comparing the pre-filled syringe (PFS) and autoinjector (AI) devices both administered to the abdomen. Bioequivalence established if both measures meet the corresponding criterion specified by the reference-scaled average bioequivalence (RSABE) approach
Time Frame: Week 8 to Week 12 dosing interval
Population: Bio-equivalence analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×µg/mL
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen
Number analyzed (Participants) | 128 | 128
h×µg/mL | 487.7 (103.5) | 474.1 (79.7)
Statistical Analysis 1: Comparison: OMB 20mg AI Abdomen vs OMB 20mg PFS Abdomen; Criteria 1 for bioequivalence testing of AUCtau; Test type: Equivalence — For reference-scaled average bioequivalence testing, both criteria have to be met: 1) geo-mean ratio needs to fall in [0.8, 1.25]; 2) 95% upper bound of the linearized criterion needs to be <= 0. This part is regarding criterion 1; Geo-mean ratio = 1.03, 90% CI 2-sided [.8 to 1.25] — The confidence interval reported in the Point Estimate section below is the one from the criterion, not the estimated confidence interval
Statistical Analysis 2: Comparison: OMB 20mg AI Abdomen vs OMB 20mg PFS Abdomen; Criteria 2 for bioequivalence testing of AUCtau; Test type: Equivalence — For reference-scaled average bioequivalence testing, both criteria have to be met: 1) geo-mean ratio needs to fall in [0.8, 1.25]; 2) 95% upper bound of the linearized criterion needs to be <= 0. This part is regarding criterion 2; 95% upper bound of the linearized criter = -.3131, 95% CI 1-sided [upper limit 0] — The upper limit reported in the Point Estimate section below is the limit on the 95% upper bound from the criterion, not the estimated upper limit of the 95% upper bound of the linearized criterion

2. Primary Outcome: Bioequivalence of 20 mg Ofatumumab Injected by Pre-filled Syringe (PFS) vs Autoinjector (AI) to Abdomen as Measured by Cmax
Description: Bioequivalence of Cmax will be measured over the time period of Week 8 to Week 12 dosing interval comparing the pre-filled syringe (PFS) and autoinjector (AI) devices both administered to the abdomen. Bioequivalence established if both measures meet the corresponding criterion specified by the reference-scaled average bioequivalence (RSABE) approach
Time Frame: Week 8 to Week 12 dosing interval
Population: Bioequivalence analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen
Number analyzed (Participants) | 128 | 128
µg/mL | 1.409 (89.2) | 1.409 (67.9)
Statistical Analysis 1: Comparison: OMB 20mg AI Abdomen vs OMB 20mg PFS Abdomen; Criteria 1 for bioequivalence testing of Cmax; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; geo-mean ratio = 1.00, 90% CI 2-sided [.8 to 1.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: OMB 20mg AI Abdomen vs OMB 20mg PFS Abdomen; Criteria 2 for bioequivalence testing of Cmax; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; 95% upper bound of the linearized criter = -0.2446, 95% CI 1-sided [upper limit 0] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Pharmacokinetics of the Study Drug as Measured by AUCtau for PFS and AI Devices When Administered to Abdomen or Thigh
Description: Pharmacokinetics following subcutaneous administration of ofatumumab to either the abdominal region or the thigh as measured by the area under the concentration-time curve over the Week 8 - Week 12 dosing interval (AUCtau)
Time Frame: Week 8 to Week 12 dosing interval
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×µg/mL
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh
Number analyzed (Participants) | 128 | 128 | 13 | 13
h×µg/mL | 487.7 (103.5) | 474.1 (79.7) | 476.0 (73.1) | 544.1 (93.8)

4. Secondary Outcome: Pharmacokinetics of the Study Drug as Measured by Cmax for PFS and AI Devices When Administered to Abdomen or Thigh
Description: Pharmacokinetics following subcutaneous administration of ofatumumab to either the abdominal region or the thigh as measured by the maximum concentration (Cmax)
Time Frame: Week 8 to Week 12 dosing interval
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh
Number analyzed (Participants) | 128 | 128 | 13 | 13
µg/mL | 1.409 (89.2) | 1.409 (67.9) | 1.563 (71.3) | 1.635 (50.7)

5. Secondary Outcome: Plasma Concentrations of the Study Drug for PFS and AI Devices When Administered to Abdomen or Thigh
Description: Plasma concentrations following subcutaneous administration of ofatumumab via PFS or AI to either the abdominal region or the thigh
Time Frame: Days 4, 7, 14, 28, 42, 56, 57, 59, 63, 70, 77, 84
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh
Number analyzed (Participants) | 128 | 130 | 13 | 13
µg/mL
  Day 4 n=128,127,13,13: number analyzed (Participants) | 128 | 127 | 13 | 13
  Day 4 n=128,127,13,13 | 0.43076 (147.591319) | 0.40075 (119.330376) | 0.86747 (24.481350) | 0.55704 (105.432315)
  Day 7 n=128, 130,13,13 | 0.33544 (133.205087) | 0.30511 (119.511321) | 0.36750 (94.007762) | 0.29662 (119.353006)
  Day 14 n=128, 130,12,11: number analyzed (Participants) | 128 | 130 | 12 | 11
  Day 14 n=128, 130,12,11 | 1.07408 (105.566707) | 0.96359 (105.735963) | 0.89788 (125.726458) | 1.30586 (83.153962)
  Day 28 Week 4 n=127, 130,13,13: number analyzed (Participants) | 127 | 130 | 13 | 13
  Day 28 Week 4 n=127, 130,13,13 | 0.95571 (113.510035) | 0.95774 (117.852822) | 1.11008 (66.780045) | 1.41434 (117.959678)
  Day 42 Week 6 n=128, 130,13,13 | 0.97327 (125.421064) | 1.12006 (113.137164) | 1.12006 (86.390639) | 1.18239 (133.082660)
  Day 56 Week 8 n=128, 130,13,13 | 0.28358 (142.760137) | 0.24644 (133.056913) | 0.23874 (98.041287) | 0.45529 (143.614763)
  Day 57 Week 8 n=127, 127,12,13: number analyzed (Participants) | 127 | 127 | 12 | 13
  Day 57 Week 8 n=127, 127,12,13 | 0.89424 (121.357310) | 0.80986 (107.929658) | 0.96356 (122.222991) | 1.04905 (54.771002)
  Day 59 Week 8 n=127, 127,13,13: number analyzed (Participants) | 127 | 127 | 13 | 13
  Day 59 Week 8 n=127, 127,13,13 | 1.24143 (103.274314) | 1.23458 (81.737063) | 1.34837 (82.596695) | 1.52705 (52.253239)
  Day 63 Week 9 n=126, 128,13,13: number analyzed (Participants) | 126 | 128 | 13 | 13
  Day 63 Week 9 n=126, 128,13,13 | 1.27031 (84.610014) | 1.23163 (77.294222) | 1.28263 (67.076249) | 1.43075 (66.345270)
  Day 70 Week 10 n=128, 127,13,13: number analyzed (Participants) | 128 | 127 | 13 | 13
  Day 70 Week 10 n=128, 127,13,13 | 0.78732 (97.440131) | 0.74111 (82.870974) | 0.67151 (82.769087) | 0.95821 (83.645358)
  Day 77 Week 11 n=127, 127,13,13: number analyzed (Participants) | 127 | 127 | 13 | 13
  Day 77 Week 11 n=127, 127,13,13 | 0.40249 (109.581877) | 0.33720 (114.373887) | 0.40173 (52.479338) | 0.54085 (97.862609)
  Early Exit n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Early Exit n=0,1,0,0 |  | 0.1870 |  |
  EOS Week 12 n=126, 118,12,13: number analyzed (Participants) | 126 | 118 | 12 | 13
  EOS Week 12 n=126, 118,12,13 | 0.20290 (113.812416) | 0.17862 (102.507484) | 0.17361 (63.899086) | 0.27276 (98.256573)

6. Secondary Outcome: Percentage of Patients With Anti-ofatumumab Antibodies
Description: Anti-drug antibodies (ADA) were assessed to evaluate the immunogenicity potential of ofatumumab. Samples for ADA assessment were taken prior to dosing at the visit. Samples were analyzed as per laboratory's SOPs by a Meso Scale Discovery (MSD) electrochemiluminescense assay. All samples confirmed to be positive for the presence of anti-ofatumumab antibodies were assessed to evaluate their ability to neutralize the ofatumumab biologic effect.
Time Frame: Baseline, Week 4, 8, 12 and Overall
Population: Safety set
Measure: Number; unit: percentage of participants
Arm/Group | OMB 20mg AI Abdomen | OMB 20mg PFS Abdomen | OMB 20mg AI Thigh | OMB 20mg PFS Thigh
Number analyzed (Participants) | 128 | 130 | 13 | 13
percentage of participants
  Baseline n= 128,130,13,13 | 0.8 | 3.1 | 0.0 | 7.7
  Week 4 n= 128,130,13,13 | 0.8 | 0.0 | 0.0 | 0.0
  Week 8 n= 124,126,13,13: number analyzed (Participants) | 124 | 126 | 13 | 13
  Week 8 n= 124,126,13,13 | 0.0 | 0.8 | 0.0 | 0.0
  Week 12 n= 125,121, 12,13: number analyzed (Participants) | 125 | 121 | 12 | 13
  Week 12 n= 125,121, 12,13 | 0.8 | 0.0 | 0.0 | 0.0
  Overall n= 128,130,13,13 | 0.8 | 3.8 | 0.0 | 7.7

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until last administration of study treatment plus 100 days post treatment, up to maximum duration of 226 days
Groups:
- OMB 20mg AI (ABD): Ofatumumab 20 mg subcutaneous (sc.) injection with autoinjector (AI) administrated on abdomen
- OMB 20mg AI (THI): Ofatumumab 20 mg subcutaneous (sc.) injection with autoinjector (AI) administrated on thigh
- OMB 20mg PFS (THI): Ofatumumab 20 mg subcutaneous (sc.) injection with pre-filled syringes (PFS) administrated on thigh
Arm/Group | OMB 20mg AI (ABD) | OMB 20mg PFS Abdomen | OMB 20mg AI (THI) | OMB 20mg PFS (THI)
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/130 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/128 | 4/130 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 61/128 | 53/130 | 7/13 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg AI (ABD) (N=128) | OMB 20mg PFS Abdomen (N=130) | OMB 20mg AI (THI) (N=13) | OMB 20mg PFS (THI) (N=13)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg AI (ABD) (N=128) | OMB 20mg PFS Abdomen (N=130) | OMB 20mg AI (THI) (N=13) | OMB 20mg PFS (THI) (N=13)
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 2 | 1 | 0 | 1
Fatigue (General disorders) | 3 | 5 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 11 | 17 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 3 | 3 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 41 | 29 | 5 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 13 | 7 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 2 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT03560739/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03560739/SAP_000.pdf